CLINICAL TRIAL: NCT00796978
Title: Safety and Efficacy of Single Agent Adjuvant Trastuzumab (Herceptin®) in Older Women With Early-Stage and Locally Advanced Breast Cancer: A Phase II Trial
Brief Title: Trastuzumab in Treating Older Women With Early-Stage Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cynthia Owusu, MD (Other)
Responsible Party: Sponsor-Investigator, Cynthia Owusu, MD, Principal Investigator, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE10107
Record Dates: First submitted 2008-11-21; First posted 2008-11-24 (Estimated); Results first posted 2020-08-03 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; HER2-positive breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Chemotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- trastuzumab (Experimental)
  Interventions: Biological: trastuzumab; Other: laboratory biomarker analysis; Procedure: adjuvant therapy; Procedure: quality-of-life assessment

INTERVENTIONS:
Biological: trastuzumab — Trastuzumab (Herceptin®) IV over 30-90 minutes on day 1. Treatment repeats every 3 weeks for up to 52 weeks in the absence of disease progression or unacceptable toxicity.
  Other Names: Herceptin
Other: laboratory biomarker analysis — Blood is collected every 6 weeks during treatment. Samples are assessed for plasma cardiac markers (N-terminal brain natriuretic protein and troponin-I) and pro-inflammatory cytokines (interleukin-6 and tumor necrosis factor-α).
Procedure: adjuvant therapy — Patients receive trastuzumab (Herceptin®) IV over 30-90 minutes on day 1. Treatment repeats every 3 weeks for up to 52 weeks in the absence of disease progression or unacceptable toxicity.
Procedure: quality-of-life assessment — Patients complete Quality of Life and Quality of Health and Comprehensive Geriatric assessments of functional, cognitive, and mental status changes at baseline, weeks 26, and 52.

SUMMARY:
RATIONALE: Monoclonal antibodies, such as trastuzumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them.

PURPOSE: This phase II trial is studying the side effects of trastuzumab and to see how well it works in treating older women with early-stage breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the 3-year cumulative incidence of cardiac events in women 60 years and older with HER2-positive breast cancer who receive single agent trastuzumab (Herceptin®) in the adjuvant setting.

Secondary

* To evaluate the 1-year cumulative incidence of asymptomatic cardiac left ventricular dysfunction in women 60 years and older with Her2-positive breast cancer who receive single agent trastuzumab in the adjuvant setting.
* To evaluate long-term cardiac toxicity (5-year cumulative incidence of cardiac events) in women 60 years and older with Her2-positive breast cancer who receive single agent trastuzumab in the adjuvant setting.
* To assess the relation between physiologic markers of chronic heart failure and trastuzumab-related cardiac dysfunction in women 60 years and older with Her2-positive breast cancer who receive single agent trastuzumab.
* To assess the relation between pro-inflammatory cytokines and trastuzumab-related cardiac dysfunction in women 60 years and older with Her2-positive breast cancer.
* To determine the effect of this drug on the health-related quality of life and functional, cognitive, and mental status of women 60 years and older with Her2-positive breast cancer.
* To determine the 5-year disease-free survival and overall survival of women 60 years and older with Her2-positive breast cancer who receive single agent trastuzumab in the adjuvant setting.

OUTLINE: This is a multicenter study.

Patients receive trastuzumab (Herceptin®) IV over 30-90 minutes on day 1. Treatment repeats every 3 weeks for up to 52 weeks in the absence of disease progression or unacceptable toxicity.

Blood is collected every 6 weeks during treatment. Samples are assessed for plasma cardiac markers (N-terminal brain natriuretic protein and troponin-I) and pro-inflammatory cytokines (interleukin-6 and tumor necrosis factor-α). Patients complete Quality of Life and Quality of Health and Comprehensive Geriatric assessments of functional, cognitive, and mental status changes at baseline, weeks 26, and 52.

After completion of study therapy, patients are followed periodically for 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the breast
* Immunohistochemical staining for Her2 protein of 3+ intensity or Her2 gene amplification of ≥ 2.0 by FISH testing.
* Life expectancy > 6 months
* ECOG performance status ≤ 2
* Node positive disease irrespective of tumor size
* Node negative disease:

  * TNM Stage (AJCC Cancer Staging Manual 6th edition) T1b-T4, N0-3, M0, irrespective of hormonal status
* Baseline LVEF ≥ lower limit of normal for a particular institution
* Complete surgical removal of invasive cancer by mastectomy or lumpectomy
* Complete staging work-up with CT of chest, abdomen, and pelvis plus bone scan or alternatively with PET scan for stage II and higher disease, or as determined by symptoms for all other stages. Additional staging work-up as per symptoms.
* Adequate bone marrow function as indicated by the following:

  * ANC >1000/µL
  * Platelets ≥100,000/µL
  * Hemoglobin >10 g/dL
* Adequate liver function, as indicated by bilirubin ≤1.5 x upper limit of normal (ULN) Adequate renal function, as indicated by creatinine ≤1.5 x ULN
* AST or ALT <2 x ULN unless related to primary disease.
* Signed informed consent

Exclusion Criteria:

* Enrollment after more than 120 days from the last day of mastectomy or lumpectomy
* Patients able to tolerate and willing to receive chemotherapy
* Prior chemotherapy for current malignancy
* Prior herceptin therapy
* Active cardiac disease

  * Myocardial infarction (asymptomatic changes on EKG suggestive of old MI is not an exclusion)
  * Angina pectoris requiring anti-anginal treatment
  * Documented congestive heart failure (CHF)
  * Current use of any therapy specifically for CHF
  * Cardiac arrhythmia requiring medication
  * Current uncontrolled hypertension (diastolic >100 mmHg or systolic > 200 mmHg)
  * Clinically significant valvular abnormality (associated with New York Heart Association (NYHA) class II, III, or IV symptoms)
  * Clinically significant pericardial effusion (associated with New York Heart Association (NYHA) class II, III, or IV symptoms)
* Past cardiac disease

  * Prior myocardial infarction (asymptomatic changes on EKG suggestive of old MI is not an exclusion)
  * Prior history of CHF
  * History of cardiomyopathy
* Other diseases and conditions

  * Evidence of metastatic breast cancer (clinical or radiological evidence)
  * Active infection
  * Concomitant malignancies or previous malignancies within the last 3 years, with the exception of adequately treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix.
  * Hypersensitivity to trastuzumab

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2009-02-05 (Actual); Primary Completion 2016-01-06 (Actual); Study Completion 2020-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Owusu, MD, MSc, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center
Locations (11):
- United States (11):
  - University of Miami, Sylvester Comprehensive Cancer Center, Miami, Florida
  - Wake Forrest, Winston-Salem, North Carolina
  - Lake/University Seidman Cancer Center, Cleveland, Ohio
  - University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - University Suburban Health Center, Cleveland, Ohio
  - UHHS Chagrin Highlands Medical Center, Cleveland, Ohio
  - Southwest General Health Center, Cleveland, Ohio
  - UHHS Westlake Medical Center, Cleveland, Ohio
  - UH-Monarch, Mayfield Heights, Ohio
  - Sharon Health Center, Wadsworth, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Trastuzumab
Started | 56
Completed | 44
Not Completed | 12
Not completed — Cardiac adverse event | 5
Not completed — Adverse Event | 4
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Population: All participants who went on study
Arm/Group | Trastuzumab
Number analyzed (Participants) | 56
Age, Customized [Count of Participants; unit: Participants]
  years: 60-69 | 19
  years: 70-79 | 23
  years: 80-89 | 13
  years: 90-99 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 55
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 49
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 56

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants Experiencing Cardiac Events at 1 Year
Description: Number of participants that experience cardiac events that include cardiac death due to congestive heart failure (CHF), Myocardial infarction (MI) or documented arrhythmia, death without definitive cause, or signs and symptoms of CHF as defined by New York Heart Association (NYHA) class III or IV symptoms.
Time Frame: At 1 year
Population: All subjects that received treatment. All related outcomes occurred within 1 year, therefore, 3-year and 5-year cumulative incidences of cardiac events and asymptomatic LV cardiac dysfunction were not performed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trastuzumab
Number analyzed (Participants) | 55
percentage of participants | 3.6 [0.09 to 13.8]

2. Secondary Outcome: Percent of Participants Experiencing Cardiac Events at 3 Years
Description: as for outcome 1
Time Frame: At 3 years
Population: Data from 3-year and 5-year echocardiograms not collected, CI of cardiac events and asymptomatic LV cardiac dysfunction were not available
Arm/Group | Trastuzumab
Number analyzed (Participants) | 0

3. Secondary Outcome: Percent of Participants Experiencing Cardiac Events at 5 Years
Description: as for outcome 1
Time Frame: At 5 years
Population: as for outcome 2
Arm/Group | Trastuzumab
Number analyzed (Participants) | 0

4. Secondary Outcome: Percent of Participants of Asymptomatic Left Ventricular (LV) Cardiac Dysfunction at 1 Year
Description: One-year cumulative incidence of LV cardiac dysfunction as measured by percent of participants that had asymptomatic LV cardiac dysfunction with/without permanent discontinuation
Time Frame: At 1 year
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Trastuzumab
Number analyzed (Participants) | 55
percent of participants | 9.1 [3.9 to 20.1]

5. Secondary Outcome: Percent of Participants With Asymptomatic LV Cardiac Dysfunction at Three Years
Description: Three-year cumulative incidence of LV cardiac dysfunction as measured by percent of participants that had asymptomatic LV cardiac dysfunction with/without permanent discontinuation
Time Frame: At 3 years
Population: as for outcome 2
Arm/Group | Trastuzumab
Number analyzed (Participants) | 0

6. Secondary Outcome: Percent of Participants With Asymptomatic LV Cardiac Dysfunction at Five Years
Description: Five-year cumulative incidence as measured by percent of participants that had asymptomatic LV cardiac dysfunction with/without permanent discontinuation
Time Frame: At 5 years
Population: as for outcome 2
Arm/Group | Trastuzumab
Number analyzed (Participants) | 0

7. Secondary Outcome: Percent of Participants With Disease-free Survival (DFS)
Description: Percent of participants with DFS measured between the time from initiation of treatment to the date of first loco-regional or distant treatment failure, ignoring any intervening contralateral breast cancers or other second primary cancers. Deaths without evidence of recurrence will be treated censoring events.
Time Frame: At 1 year
Population: All participants that received treatment.
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Trastuzumab
Number analyzed (Participants) | 55
Percent of participants | 96.36 [86.23 to 99.08]

8. Secondary Outcome: Percent of Participants With DFS
Description: as for outcome 7
Time Frame: At 2 years
Population: All participants that received treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trastuzumab
Number analyzed (Participants) | 55
percentage of participants | 94.47 [83.83 to 98.18]

9. Secondary Outcome: Percent of Participants With Disease-free Survival (DFS)
Description: as for outcome 7
Time Frame: At 3 years
Population: All participants that received treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trastuzumab
Number analyzed (Participants) | 55
percentage of participants | 92.46 [81.13 to 97.11]

10. Secondary Outcome: Percent of Participants With Disease-free Survival (DFS)
Description: as for outcome 7
Time Frame: At 5 years
Population: All participants that received treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trastuzumab
Number analyzed (Participants) | 55
percentage of participants | 86.4 [73.59 to 93.30]

11. Secondary Outcome: Overall Survival (OS) as Measured by Percent of Participants Alive at 1 Year
Description: OS defined as percent of participants alive between time from initiation of treatment to the date of protocol-defined outcome from any cause and censored to the date of last follow-up for survivors.
Time Frame: Up to 1 years
Population: All participants that received treatment.
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Trastuzumab
Number analyzed (Participants) | 55
percent of participants | 100.0 [100.0 to 100.0]

12. Secondary Outcome: Overall Survival (OS) as Measured by Percent of Participants Alive at 2 Years
Description: as for outcome 11
Time Frame: Up to 2 years
Population: All participants that received treatment.
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Trastuzumab
Number analyzed (Participants) | 55
percent of participants | 100.0 [100.0 to 100.0]

13. Secondary Outcome: Overall Survival (OS) as Measured by Percent of Participants Alive at 3 Years
Description: as for outcome 11
Time Frame: Up to 3 years
Population: All participants that received treatment.
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Trastuzumab
Number analyzed (Participants) | 55
percent of participants | 94.23 [83.17 to 98.10]

14. Secondary Outcome: Overall Survival (OS) as Measured by Percent of Participants Alive at 5 Years
Description: as for outcome 11
Time Frame: Up to 5 years
Population: All participants that received treatment.
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Trastuzumab
Number analyzed (Participants) | 55
percent of participants | 90.2 [79.91 to 97.70]

15. Secondary Outcome: Mean Change in Quality of Life From Baseline to Mid-treatment
Description: Quality of life was assessed by using the mean change in Functional Assessment of Cancer Therapy-Breast (FACTB) scoring instrument. The Functional Assessment of Cancer Therapy-Breast (FACT-B) is a 37-item instrument designed to measure five domains of HRQOL in breast cancer patients: Physical, social, emotional, and functional well-being, as well as a breast-cancer subscale (BCS). Each question response is based on a 5-point Likert-type scale. Scores range from 0-148. High scores indicate better QOL.
Time Frame: From Baseline to mid-treatment (week 26)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Trastuzumab
Number analyzed (Participants) | 33
score on a scale | -2.8 (17.9)

16. Secondary Outcome: Mean Change in Quality of Life From Baseline to End of Treatment
Description: as for outcome 15
Time Frame: From baseline to end-of-treatment (52 weeks)
Population: Only participants with no missing values at baseline and mid-treatment and at baseline and end of treatment were included
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Trastuzumab
Number analyzed (Participants) | 18
score on a scale | -9.2 (24.3)

17. Secondary Outcome: Mean Change in Functional Status
Description: Mean Change in ADL/IADL scores From Baseline to Mid-treatment. The functional status will be measured by a Comprehensive Geriatric Assessment comprised of two validated instruments: Katz's Activity of Daily Living (ADL) instrument and Lawton's Instrumental of Activities of Daily Living (IADL). The IADL scale contains eight items with a summary score from 0 (low function) to 8 (high function), with higher scores indicating higher function. The ADL scale contains six items with a summary score of 0 to 6, with higher scores indicating higher independence. A score of 6 indicates complete independence; a score of 4 indicates moderate impairment; 2 or less indicates severe functional impairment. The scores of both scales will be added together for a comprehensive geriatric assessment score.
Time Frame: From Baseline to mid-treatment (week 26)
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Trastuzumab
Number analyzed (Participants) | 41
score on a scale | -0.05 (0.74)

18. Secondary Outcome: Mean Change in Functional Status
Description: Mean Change in ADL/IADL scores From Baseline to End of Treatment. The functional status will be measured by a Comprehensive Geriatric Assessment comprised of two validated instruments: Katz's Activity of Daily Living (ADL) instrument and Lawton's Instrumental of Activities of Daily Living (IADL). The IADL scale contains eight items with a summary score from 0 (low function) to 8 (high function), with higher scores indicating higher function. The ADL scale contains six items with a summary score of 0 to 6, with higher scores indicating higher independence. A score of 6 indicates complete independence; a score of 4 indicates moderate impairment; 2 or less indicates severe functional impairment. The scores of both scales will be added together for a comprehensive geriatric assessment score.
Time Frame: baseline to end-of-treatment (52 weeks)
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Trastuzumab
Number analyzed (Participants) | 31
score on a scale | -0.26 (1.15)

19. Secondary Outcome: Mean Change in Cognitive Status
Description: Mean Change in Mini Mental Status Exam (MMSE scores) From Baseline to Mid-treatment. The Mini-Mental Status Exam contains 11 items to gauge cognitive function. The minimum score is 0. The maximum score is 30. A score of 23 or lower is indicative of cognitive impairment. The higher the score, the better the participant's function (Scores 30-24 indicate uncertain cognitive impairment; scores 23-18 indicate mild to moderate cognitive impairment; scores 17-0 indicate severe cognitive impairment).
Time Frame: From Baseline to mid-treatment (week 26)
Population: Only participants with no missing values at baseline and mid treatment and at baseine and end of treatment were included
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Trastuzumab
Number analyzed (Participants) | 40
score on a scale | 0 (1.94)

20. Secondary Outcome: Mean Change in Cognitive Status
Description: Mean Change in Mini Mental Status Exam (MMSE scores) From Baseline to End of Treatment. The Mini-Mental Status Exam contains 11 items to gauge cognitive function. The minimum score is 0. The maximum score is 30. A score of 23 or lower is indicative of cognitive impairment. The higher the score, the better the participant's function (Scores 30-24 indicate uncertain cognitive impairment; scores 23-18 indicate mild to moderate cognitive impairment; scores 17-0 indicate severe cognitive impairment).
Time Frame: From baseline to end-of-treatment (52 weeks)
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Trastuzumab
Number analyzed (Participants) | 29
score on a scale | -0.59 (1.15)

21. Secondary Outcome: Mean Change in Psychosocial Status (Depression)
Description: Mean Change in Geriatric Depression Scores From Baseline to Mid-treatment. The Geriatric Depression Scale (GDS) is a validated tool with 15 items. The minimum score is 0, and the maximum is 15. Scores of 0-4 are considered normal, depending on age, education, and complaints; 5-8 indicate mild depression; 9-11 indicate moderate depression; and 12-15 indicate severe depression.
Time Frame: From Baseline to mid-treatment (week 26)
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Trastuzumab
Number analyzed (Participants) | 39
score on a scale | 0.15 (1.60)

22. Secondary Outcome: Mean Change in Psychosocial Status (Depression)
Description: Mean Change in Geriatric Depression Scores from Baseline to End of Treatment. The Geriatric Depression Scale (GDS) is a validated tool with 15 items. The minimum score is 0, and the maximum is 15. Scores of 0-4 are considered normal, depending on age, education, and complaints; 5-8 indicate mild depression; 9-11 indicate moderate depression; and 12-15 indicate severe depression.
Time Frame: From baseline to end-of-treatment (52 weeks)
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Trastuzumab
Number analyzed (Participants) | 28
score on a scale | -0.39 (1.83)

23. Secondary Outcome: Mean Change in Psychosocial Status (Social Support)
Description: Mean Change in MOS social support scores From Baseline to Mid-treatment. The Medical Outcomes Study (MOS) Social Support survey tool measures multiple domains. It is a 19-item tool comprised of four subscales in one overall summary index. The subscales are Emotional/Informational Support, Tangible Support, Affectionate support, and Positive Social Interaction. The overall index score is determined by calculating the mean of all 19 items. Scores range from 19 to 95, with higher scores indicating high support availability to participants.
Time Frame: From Baseline to mid-treatment (week 26)
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Trastuzumab
Number analyzed (Participants) | 37
score on a scale | -1.03 (22.4)

24. Secondary Outcome: Mean Change in Psychosocial Status (Social Support)
Description: Mean Change in MOS social support scores From Baseline to End of Treatment. The Medical Outcomes Study (MOS) Social Support survey tool measures multiple domains. It is a 19-item tool comprised of four subscales in one overall summary index. The subscales are Emotional/Informational Support, Tangible Support, Affectionate support, and Positive Social Interaction. The overall index score is determined by calculating the mean of all 19 items. Scores range from 19 to 95, with higher scores indicating high support availability to participants.
Time Frame: From baseline to end-of-treatment (52 weeks)
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Trastuzumab
Number analyzed (Participants) | 28
score on a scale | -7.53 (22.12)

25. Secondary Outcome: Mean Change in Nutritional Status
Description: Mean Change in Mini Nutrition Assessment scores From Baseline to Mid-treatment. The Mini Nutritional Screening is a scale comprised of six questions. The sum of the six questions is totaled to determine a score which is designed to assess if there is a risk of malnutrition. The highest score possible, 14, indicated no risk, and the minimum score of 0 indicates the highest risk possible. 12 points or greater is considered no risk or normal. Meanwhile, a score below 11 indicates possible malnutrition.
Time Frame: From Baseline to mid-treatment (week 26)
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Trastuzumab
Number analyzed (Participants) | 38
score on a scale | 0.14 (2.11)

26. Secondary Outcome: Mean Change in Nutritional Status
Description: Mean Change in Mini Nutrition Assessment scores From Baseline to End of Treatment. The Mini Nutritional Screening is a scale comprised of six questions. The sum of the six questions is totaled to determine a score which is designed to assess if there is a risk of malnutrition. The highest score possible, 14, indicated no risk, and the minimum score of 0 indicates the highest risk possible. 12 points or greater is considered no risk or normal. Meanwhile, a score below 11 indicates possible malnutrition.
Time Frame: From baseline to end-of-treatment (52 weeks)
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Trastuzumab
Number analyzed (Participants) | 22
score on a scale | -0.39 (2.47)

27. Secondary Outcome: Mean Change in Pro-inflammatory Cytokines
Description: Mean change in pro-inflammatory cytokines from baseline to mid-treatment
Time Frame: From Baseline to mid-treatment (week 26)
Population: Analysis was not completed due to too many missing values that affected the validity of results and interpretation of data.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Trastuzumab
Number analyzed (Participants) | 45
pg/ml | NA (NA) — Analysis was not completed due to too many missing values that affected the validity of results and interpretation of data.

28. Secondary Outcome: Mean Change in Pro-inflammatory Cytokines
Description: Mean change in pro-inflammatory cytokines from baseline to end of treatment
Time Frame: From baseline to end-of-treatment (52 weeks)
Population: Unable to complete analysis due to too many missing values that affected the validity of results and interpretation of data.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Trastuzumab
Number analyzed (Participants) | 45
pg/ml | NA (NA) — Unable to complete analysis due to too many missing values that affected the validity of results and interpretation of data.

29. Secondary Outcome: Mean Change in Plasma Cardiac Markers
Description: Mean change in plasma cardiac markers from baseline to mid-treatment
Time Frame: From Baseline to mid-treatment (week 26)
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Trastuzumab
Number analyzed (Participants) | 24
pg/ml | NA (NA) — Unable to complete analysis due to too many missing values that affected the validity of results and interpretation of data.

30. Secondary Outcome: Mean Change in Plasma Cardiac Markers
Description: Mean change in plasma cardiac markers from baseline end of treatment
Time Frame: From baseline to end-of-treatment (52 weeks)
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Trastuzumab
Number analyzed (Participants) | 24
pg/ml | NA (NA) — Unable to complete analysis ue to too many missing values that affected the validity of results and interpretation of data.

ADVERSE EVENTS:
Time Frame: Adverse Event Data was collected up to 5 years of study participation.
Arm/Group | Trastuzumab
All-Cause Mortality (participants affected / at risk) | 5/56
Serious Adverse Events (participants affected / at risk) | 8/56
Other Adverse Events (participants affected / at risk) | 17/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trastuzumab (N=56)
Heart failure (Cardiac disorders) | 1 (3)
Dehydration (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils - Bladder (urinary) (Infections and infestations) | 1 (1)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1 (2)
Fracture (Musculoskeletal and connective tissue disorders) | 2 (2)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary/Upper Respiratory - Other (Specify, _Flu_) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1)
Platelets (Blood and lymphatic system disorders) | 1 (1)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trastuzumab (N=56)
Hypertension (Cardiac disorders) | 6 (7)
Left ventricular systolic dysfunction (Cardiac disorders) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 2 (3)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Infection with unknown ANC - Urinary tract NOS (Infections and infestations) | 1 (1)
Glomerular filtration rate (Metabolism and nutrition disorders) | 1 (2)
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 1 (1)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1 (2)
Left ankle sprain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain- Buttock (Musculoskeletal and connective tissue disorders) | 1 (1)
CNS cerebrovascular ischemia (Nervous system disorders) | 1 (1)
Confusion (Nervous system disorders) | 1 (1)
Pain-Kidney (General disorders) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-12-28): https://cdn.clinicaltrials.gov/large-docs/78/NCT00796978/Prot_SAP_000.pdf
  • Informed Consent Form (2022-05-26): https://cdn.clinicaltrials.gov/large-docs/78/NCT00796978/ICF_002.pdf